CLINICAL TRIAL: NCT02820571
Title: The Oxford Pain, Activity and Lifestyle (OPAL) Cohort Study
Acronym: OPAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID: 196643
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The OPAL study is about health outcomes in older adults. The investigators are surveying 4,000 adults across England to see how health and physical activity change over time. The information that is collected will help the investigators to understand how a person's health, including conditions such as back pain, affect their mobility as they age, and provide insight into improving the management of health in older adults.

DETAILED DESCRIPTION:
The Oxford Pain, Activity and Lifestyle (OPAL) study is a large cohort study of community dwelling adults (n=4000) aged 65 years and over. This cohort data will allow the investigators to describe the prevalence, severity, course and prognosis a range of musculoskeletal problems in older people. The initial focus is to evaluate the impact of back pain on important health outcomes for older people (quality of life, mobility, falls and fractures). In order to do this, the investigators will study people with and without back pain at the inception of the cohort. The OPAL cohort will be followed for 5 years in the first instance and the investigators will study a range of factors hypothesised to moderate and mediate the effects of back and other musculoskeletal pain for example, co-morbidities.

The OPAL cohort will be sampled from older people registered with primary care practices.

The investigators aim to develop a prognostic tool using the cohort data that will help older people, GPs and other health professionals identify when LBP is a risk factor for disability, functional limitation and loss of mobility, and when LBP should be prioritised as a treatment target.

ELIGIBILITY:
Inclusion Criteria:

* Registered with a primary care practice.
* 65 years and over.

Exclusion Criteria:

* Living in a residential care or nursing home.
* Has a terminal condition with a life expectancy of less than 6 months.
* Any substantial health or social concern that, in the opinion of the patient's GP, would place the patient at increased risk or inability to participate including known inability to provide informed consent e.g. Dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants in the OPAL cohort study will be community dwelling adults, aged 65 years and over, registered with a primary care practice
Sampling Method: Probability Sample
Enrollment: 5409 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Life-Space assessment | 5 years
  Life-Space Assessment measures mobility in terms of the spatial extent of a person's life. The purpose of the Life-Space Assessment is to determine a person's usual pattern of mobility during the month preceding the assessment. Life-space is defined based upon the distance a person routinely travels to perform activities over this time frame. This includes determining how far and how often the person leaves his or her place of residence and the degree of independence the person has.
Self-reported falls | 5 years
  The investigators will use the definitions of the Prevention of Falls Network Europe consensus on core outcomes which provides standard definitions of falls.
EQ-5D-5L | 5 years
  Disability and health-related quality of life is measured by the EQ-5D-5L
Tilburg Frailty Indicator | 5 years
Health Resource Use | 5 years
  Health resource use will be captured through routine health service data collection systems (Hospital Episode Statistics: inpatient, accident and emergency and diagnostic imaging datasets).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lamb, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Botnar Research Centre, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Lyle S, Williamson E, Darton F, Griffiths F, Lamb SE. A qualitative study of older people's experience of living with neurogenic claudication to inform the development of a physiotherapy intervention. Disabil Rehabil. 2017 May;39(10):1009-1017. doi: 10.1080/09638288.2016.1177611. Epub 2016 May 23. PMID 27216498